CLINICAL TRIAL: NCT03662126
Title: A Phase 2/3 Randomized, Controlled, Open-Label Study of KRT 232 in Subjects With Primary Myelofibrosis (PMF), Post Polycythemia Vera MF (Post-PV-MF), Or Post Essential Thrombocythemia MF (Post-ET-MF) Who Are Relapsed or Refractory to Janus Kinase (JAK) Inhibitor Treatment
Brief Title: KRT-232 Versus Best Available Therapy for the Treatment of Subjects With Myelofibrosis Who Are Relapsed or Refractory to JAK Inhibitor Treatment
Acronym: BOREAS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KRT-232-101
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Primary Myelofibrosis (PMF); Post-Polycythemia Vera MF (Post-PV-MF); Post-Essential Thrombocythemia MF (Post-ET-MF)
Keywords: navtemadlin
MeSH Terms: conditions — Primary Myelofibrosis | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part A Cohort 1 (Experimental): KRT-232 120 mg by mouth once daily for Days 1-7, off treatment for Days 8-21 (21-day cycles)
  Interventions: Drug: KRT-232
- Part A Cohort 2 (Experimental): KRT-232 240 mg by mouth once daily for Days 1-7, off treatment for Days 8-21 (21-day cycles)
  Interventions: Drug: KRT-232
- Part A Cohort 3 (Experimental): KRT-232 240 mg by mouth once daily for Days 1-7, off treatment for Days 8-28 (28-day cycles)
  Interventions: Drug: KRT-232
- Part A Cohort 4b (Experimental): KRT-232 240 mg by mouth once daily for Days 1-5, off treatment for Days 6-28 (28-day cycles)
  Interventions: Drug: KRT-232
- Part B Arm 1 KRT-232 (Experimental): KRT-232 240 mg by mouth once daily for Days 1-7, off treatment for Days 8-28 (28-day cycles)
  Interventions: Drug: KRT-232
- Part B Arm 2 Best Available Therapy (Active Comparator): Best available therapy at the discretion of the investigator, on a 28-day cycle.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: KRT-232 — KRT-232, administered by mouth
  Arms: Part A Cohort 1; Part A Cohort 2; Part A Cohort 3; Part A Cohort 4b; Part B Arm 1 KRT-232
Drug: Best Available Therapy (BAT) — Best available therapy options include:
  1. hydroxyurea
  2. chemotherapy or
  3. supportive care (including but not limited to corticosteroids and androgens; JAK inhibitors not allowed).
  Arms: Part B Arm 2 Best Available Therapy

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, for the treatment of patients with myelofibrosis (MF) who no longer benefit from treatment with a JAK inhibitor. Inhibition of MDM2 is a novel mechanism of action in MF.

This study will be conducted in 2 phases. Phase 2 will determine the KRT-232 recommended dose and dosing schedule; Phase 3 will test KRT-232 vs Best Available Therapy (BAT). Patients in the Phase 3 part of the study will be randomized 2:1 to receive either KRT-232 (Arm 1) or BAT (Arm 2). The BAT administered will be determined by the treating physician, with the option to "cross-over" to KRT-232 treatment after 6 months of BAT or if the disease worsens at any time.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PMF, post-PV MF or post-ET MF (WHO)
* High, intermediate-2, or intermediate-1 risk Dynamic International Prognostic System (DIPSS)
* Failure of prior treatment with JAK inhibitor
* ECOG ≤ 2

Exclusion Criteria:

* Prior splenectomy
* Splenic irradiation within 3 months prior to randomization
* History of major hemorrhage or intracranial hemorrhage within 6 months prior to randomization
* History of stroke, reversible ischemic neurological defect or transient ischemic attack within 6 months prior to randomization
* Prior MDM2 inhibitor therapy or p53-directed therapy
* Prior allogeneic stem-cell transplant or plans for allogeneic stem cell transplant
* History of major organ transplant
* Grade 2 or higher QTc prolongation (> 480 milliseconds per NCI-CTCAE criteria, version 5.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
(Part A Only) Spleen Volume Reduction (SVR) | 24 weeks
  The proportion of subjects achieving a ≥ 35% spleen volume reduction (SVR) from Baseline to Week 24, as assessed by magnetic resonance imaging (MRI) or computed tomography (CT) scan
(Part B Only) Spleen Volume Reduction (SVR) | 24 Weeks
  The proportion of subjects achieving SVR of ≥ 35% at Week 24 by MRI/CT scan (central review)

SECONDARY OUTCOMES:
(Part A only) Improvement in Total Symptom Score (TSS) | 48 weeks
  The proportion of subjects who have at least a 50% reduction from Baseline to Week 24 and Week 48 in the total symptom score as measured by the modified MPN-SAF v2.0
(Part B only) Improvement of Total Symptom Score (TSS) | 24 Weeks
  The proportion of subjects who have at least a 50% reduction from Baseline to Week 24 in the total symptom score as measured by the MF-SAF v4.0
(Part B only) Overall Survival (OS) | 48 months
  Time from randomization to death from any cause
(Part B only) Progression free survival (PFS) | 48 months
  Time from randomization to either first occurrence of disease progression or death due to any cause
(Part B Only) Overall Spleen Volume Reduction (SVR) | 48 months
  The proportion of subjects in each arm achieving SVR of ≥ 35% at any time by MRI/CT scan (central review)
(Part B Only) Spleen Response Duration | 48 months
  Time from initial SVR of ≥ 35% by MRI/CT (central review) until the first occurrence of disease progression
(Part B Only) Rate of conversion from RBC transfusion dependent to independent | 24 weeks
  The proportion of subjects who have RBC transfusion independence at week 24

CONTACTS AND LOCATIONS:
Locations (191):
- United States (19):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Center - Palo Alto, Stanford, California
  - Innovative Clinical Research Institute, Whittier, California
  - University Cancer Institute, Boynton Beach, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - New York Presbyterian/Weill Cornell Medical Center, New York, New York
  - Mt. Sinai, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (4):
  - Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Instituto Medico Alexander Fleming, Buenos Aires
  - Centro Medico San Luis, CABA
  - Hospital Privado - Centro Medico de Cordoba - Oncology, Córdoba
- Australia (6):
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hosital, Murdoch, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - The Alfred Hospital, Melbourne
  - South Eastern Private Hospital, Noble Park
  - Icon Cancer Center, South Brisbane
- Brazil (12):
  - Centro de oncologia Leonardo da Vinci, Fortaleza, Ceará
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - UNICAMP - Universidade Estadual de Campinas Hemocentro, Campinas, São Paulo
  - Hospital das Clínicas UFG, Goiânia
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital de Clinicas de Porto Alegre - Centro de Pesquisa Clinica, Porto Alegre
  - Associação Educadora São Carlos AESC - Hospital Mãe de Deus - Centro de Pesquisa, Porto Alegre
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Hospital A C Camargo - Fundacao Antonio Prudente, São Paulo
  - Instituto D'or de Pesquisa e Ensino, São Paulo
  - Hospital das Clínicas da Universidade de São Paulo, São Paulo
  - Instituto COI São Paulo, São Paulo
- Bulgaria (7):
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski, Pleven, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Georgi, Plovdiv, Plovdiv
  - Military Medical Academy, Multiprofile for active treatment, Sofia, Sofia
  - Acibadem City Clinic Tokuda Hospital, Sofia, Sofia
  - Specialized Hospital for Active Therapy of Hematological Disorders, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska, Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment Saint Ivan Rilski, Sofia, Sofia
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Croatia (3):
  - General Hospital Sibenik, Šibenik
  - Clinical Hospital Centre Osijek, Zagreb
  - KB Sestre Milosrdnice, Zagreb
- Czechia (3):
  - FN Hradec Kralove, Králová
  - Vseonecma fakultni nemocrince V Praze, New Town
  - Fakultní Nemocnice Olomouc, Olomouc
- France (11):
  - Centre Hospitalier Universitaire D'Amiens (Hopital Sud) - Hématologie Clinique, Amiens
  - Center Hospitalier Universitaire d'Angers, Angers
  - C.H de la Côte Basque - Serviv, Bayonne
  - Centre Hospitalier Regional Universitaire Brest Hopital Morvan, Brest
  - Centre Hospitalier Universitaire of Caen Normandie - Côte de Nacre, Caen
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Hopital Paul Brousse - Aphp Hôpitaux Universitaires Paris Su, Villejuif
- Germany (12):
  - Klinikum Rechts der Isar der Technischen Universität München Apotheke, München, Bavaria
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Gemeinschaftspraxis Haematologie - Onkologie - Hauptstelle, Dresden, Saxony
  - Technische Universität Dresden, Dresden, Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - UKE - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Praxis für Hämatologie und Onkologie, Saarbrücken
- Greece (3):
  - University General Hospital of Ioannina, Ioannina, Ioannina
  - University Campus of Patras - Hematology, Pátrai
  - AHEPA General Hospital of Thessaloniki, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital - Medicine, Shatin
- Hungary (7):
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Markusovszky Egyetemi Oktatókórház, Szombathely, Vas County
  - Semmelweis Egyetem, Budapest
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum, Debrecen
  - Szegedi Tudományegyetem, Szeged
- Israel (11):
  - Ha'Emek Medical Center, Afula
  - Assuta Ashdod University Hospital, Ashdod
  - Rambam Medical Centre, Haifa
  - Carmel MC, Haifa
  - Hadassah Medical Organisation, Jerusalem
  - Hematology Institute, Kfar Saba
  - Western Galilee Hospital - Nahariya, Nahariya
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center - Oncology, Tel Aviv
  - Assuta MC, Tel Aviv
  - Assaf Harofeh Medical Center - Hematology, Ẕerifin
- Italy (15):
  - A.O. San Gerardo di Monza - L'Ospedale San Gerardo di Monza e l'Università di Milano, Monza, Lombardy
  - PO Civile SS.Antonio e Biagio, Alessandria
  - AOU Ospedali Riuniti Umberto I G.M. Lancisi G. Salesi, Ancona
  - A.O.di Bologna Policl.S.Orsola, Bologna
  - AO Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Policlinico - Vittorio Emanuele, Catania
  - AOU Careggi, Florence
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST IRCCS, Meldola
  - Ospedale Maggiore Policlinico, Fondazione IRCCS Ca' Granda, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Maggiore della Carità, Novara
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord - Pesaro, Pesaro
  - Arcispedale S. Maria Nuova, AO di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Agostino Gemelli, Roma
  - A.O. Citta della Salute e della Scienza di Torino, Torino
- Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas, Lithuania
- Mexico (4):
  - Universidad Autonoma de Nuevo Leon (UANL) - Hospital Universitario "Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Instituto Mexicano del Seguro Social, Monterrey
  - Oaxaca Site Management Organization OSMO, Oaxaca City
  - Sociedad de Metabolismo y Corazón S.C. - Oncology, Veracruz
- Philippines (2):
  - Perpetual Succour Hospital - Hemat/Transfusion Med, Cebu City
  - University of the Philippines - Philippine General Hospital, Manila
- Poland (9):
  - Dolnośląskie Centrum Transplantacji Komórkowych z Krajowym Bankiem Dawców Szpiku, Wroclaw, Lower Silesian Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów, Podkarpackie Voivodeship
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Zespół Szpitali Miejskich, Chorzów, Silesian Voivodeship
  - Szpital Uniwersytecki nr 2 im dr. Jana Biziela, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - SPZOZ MSWiA z Warminsko - Mazurskim Centrum Onkologii, Olsztyn
  - Szpital Wojewódzki w Opolu, Opole
  - Clinical Research Center Spółka z Ograniczoną Odpowiedzialnością Medic-R sp. k., Poznan
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk
- Portugal (5):
  - H. Infante Dom Pedro. Centro Hospitalar do Baixo Vouga, Aveiro
  - Hospital de Braga, Braga
  - Instituto Português de Oncologia de Coimbra, Coimbra
  - Champalimaud Cancer Center, Lisbon
  - H. São Francisco Xavier-Centro Hospitalar Lisboa Ocidental, Lisbon
- Romania (10):
  - Cen Med de Diagn si Trat Amb NEOMED, Brasov
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Medicover, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Tg Mures, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
  - Oncomed, Timișoara
- Russia (3):
  - Clinical oncological dispensary, Omsk
  - Saint-Petersburg SMU I.P.Pavlov, Saint Petersburg
  - Oncologic dispensary of Komi Republic, Syktyvkar
- South Korea (8):
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra - H. de Navarra, Hematología C/ de Irunlarrea, 3, Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Doctor Peset, Valencia
  - H. Quirón Zaragoza, Zaragoza
- Taiwan (4):
  - National Taiwan University Hospital, Taipei City, Taipei
  - Chang Gung Medical Foundation - ChiaYi Chang Gung Memorial Hospital - Chiayi Branch, Chiayi City
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
- Thailand (5):
  - Ramathibodi Hospital - Mahidol University - Hematology, Bangkok
  - Siriraj Hospital, Bangkok
  - Thammasat University Hospital, Khlong Luang
  - Srinagarind Hospital (KhonKaen University), Khon Kaen
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (8):
  - Sakarya Research and Training Hospital, Adapazarı
  - Ankara University Faculty of Medicine, Ankara
  - Gazi University Medical Faculty, Ankara
  - Pamukkale University, Denizli
  - Gaziantep University Faculty of Medicine, Gaziantep
  - Inonu University Turgut Ozal Medical Center, Malatya
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis University Medical Faculty - Hematology, Samsun
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - NHS Greater Glasgow and Clyde, Glasgow
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

REFERENCES:
- [Background] Al-Ali, H.K.; Delgado, R.G.; Lange, A.; Pluta, A.; McLornan, D.; Vachhani, P.; Damaj, G.L.; Jost, P.J.; Rejto, L.; Hus, M.; et al. KRT-232, A First-In-Class, Murine Double Minute 2 Inhibitor, for Myelofibrosis Relapsed or Refractory to Janus-Associated Kinase Inhibitor Treatment. Eha. Libr. 2020, 295035, S215